CLINICAL TRIAL: NCT04179526
Title: The Efficacy and Mechanisms of Change of a Transdiagnostic Internet-delivered REBT Intervention for Adolescents With Internalizing Problems: A Randomized Controlled Trial
Brief Title: Transdiagnostic Internet-delivered REBT Intervention for Adolescents' Internalizing Problems
Acronym: REBTonAd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Babes-Bolyai University (Other)
Responsible Party: Principal Investigator, Anca Dobrean, Professor, Babes-Bolyai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PN-III-P4-ID-PCE-2016-0861
Record Dates: First submitted 2019-11-14; First posted 2019-11-27 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Anxiety Disorders; Social Anxiety Disorder; Generalized Anxiety Disorder; Panic Disorder; Persistent Depressive Disorder; Major Depressive Disorder
Keywords: transdiagnostic; anxiety; depression; REBT; adolescents; Internet intervention
MeSH Terms: conditions — Anxiety Disorders; Phobia, Social; Generalized Anxiety Disorder; Panic Disorder; Depressive Disorder, Major; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transdiagnostic Internet-delivered REBT (Experimental): Protocol is based on Rational Emotive Therapy (Ellis, 1962, 1994), structured in 8 modules delivered over 6 weeks (Module 1- Introduction and psychoeducation about emotions, Module 2 - Psychoeducation anxiety and depression, Module 3 - Relaxation, Module 4 - Negative patterns of thinking and cognitive restructuring, Module 5 - Problem solving, Module 6 - Exposure and Behavioral activation, Module 7 - Positive emotions and Module 8 - Gaining maintenance)
  Interventions: Behavioral: Transdiagnostic Internet-delivered REBT
- Waitlist (No Intervention): Participants in the control group will complete pre-treatment and post-treatment assessments. After participants in the experimental group complete post-treatment assessment, they will receive the intervention.

INTERVENTIONS:
Behavioral: Transdiagnostic Internet-delivered REBT — The protocol is based on Rational Emotive and Behavioral Therapy (REBT; Ellis, 1962, 1994). The program will consist of 8 modules, delivered online over six weeks.
  Arms: Transdiagnostic Internet-delivered REBT

SUMMARY:
To investigate the efficacy and mechanisms of change of an Internet-delivered transdiagnostic REBT intervention for adolescents with internalizing problems.

DETAILED DESCRIPTION:
The main objectives of this study are to evaluate the efficacy and mechanisms of change of an Internet-delivered Rational Emotive Behavior Therapy for adolescents (12-15 years) diagnosed with a principal anxiety or depressive disorder according to DSM-5 criteria. Participants will be randomly allocated to one of the two groups: experimental (REBTonAd) and waitlist control. The intervention is structured in 8 modules and will be delivered over six weeks. Assessments will be conducted at four time points: baseline, post-treatment, 3-month follow-up, and 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 12 and 15 years
* A principal diagnosis of Social Anxiety Disorder, Generalized Anxiety Disorder, Panic Disorder, Persistent Depressive Disorder, or Major Depressive Disorder as defined by DSM-5 (APA, 2013)
* Not currently following another treatment (psychotherapy, pharmacological treatment);
* Internet access
* Ability to read and write Romanian

Exclusion Criteria:

* Suicidal ideation
* Severe depression
* Any physical and mental health acute problem that requires hospitalization
* Diagnosed with autism spectrum disorder, psychosis, bipolar disorder or mental disability

Ages: 12 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2020-01-25 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Internalizing problems measured with the Youth Self-Report 11/18 (YSR; Achenbach & Rescorla, 2001) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in self-reported internalizing problems from baseline to post-treatment, at 6 months post treatment. Higher scores indicate higher levels of internalizing problems.

SECONDARY OUTCOMES:
Automatic Thoughts QuestionnaireShort Version (ATQ-SV; Netemeyer et al., 2002) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in negative automatic thoughts from baseline. Higher scores indicating higher levels of negative automatic thoughts.
The child and adolescent scale of irrationality (CASI; Bernard & Cronan, 1999) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in irrational beliefs from baseline. Higher scores indicate higher levels of irrational beliefs.
The Questionnaire for Measuring Health-Related Quality of Life in Children and Adolescents, The Revised Version - adolescent version (Kiddo-KINDL; Ravens-Sieberer, & Bullinger, 1998) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in quality of life from baseline from baseline. Higher scores indicate higher levels of quality of life.
The Adolescent Peer Relations Instrument (APRI; Parada, 2000) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in bullying victimization from baseline. Higher scores indicate higher levels of peer victimization.
Principal diagnosis based on Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria | Baseline, 6-month follow-up
  Diagnostic interview for anxiety disorders and/or depressive disorders

OTHER OUTCOMES:
The anxiety subscale from The Beck Youth Inventories™ -Second Edition for Children and Adolescents (Beck, Beck, & Jolly, 2005). | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in anxiety subscale from baseline. This subscale contains 20 items, rated on a 4 point Likert scale, with 0 = Never and 3 = Always. The total score is obtained by summing the 20 items, with higher scores indicating higher symptoms of anxiety.
The depression subscale from the Beck Youth Inventories™ -Second Edition for Children and Adolescents (Beck et al., 2005) | Baseline, Immediately after the intervention (an expected average of 6 weeks), 6-month follow-up
  Change in depression subscale from baseline. This subscale contains 20 items, rated on a 4 point Likert scale, with 0 = Never and 3 = Always. The total score is obtained by summing the 20 items, with higher scores indicating higher symptoms of depression.
Client Satisfaction Scale | Immediately after the intervention (an expected average of 6 weeks)
  Satisfaction with the program. Higher scores indicate higher treatment satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Anca Dobrean, Ph.D., Principal Investigator — Babeș-Bolyai University
Locations (1):
- Babeș-Bolyai University, Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dobrean A, Poetar CR, Florean IS, Balan R, Andersson G. Transdiagnostic Internet-delivered intervention for children and adolescents with anxiety and depressive disorders: a randomized controlled trial. NPJ Digit Med. 2026 Jan 16. doi: 10.1038/s41746-026-02341-x. Online ahead of print. PMID 41545507